CLINICAL TRIAL: NCT01793441
Title: A Multi-Center, Randomized, Double-Blind, 12-Week, Parallel Group, Placebo-Controlled Proof of Concept Study to Investigate the Efficacy and Safety of RG7314 in Individuals With Autism Spectrum Disorders (ASD)
Brief Title: A Study of RG7314 to Investigate Efficacy and Safety in Individuals With Autism Spectrum Disorders (ASD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP28420; 2012-005597-55 (EudraCT Number)
Record Dates: First submitted 2013-02-14; First posted 2013-02-15 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive placebo matching to RG7314 in each stage (Stage I, II, III and IV) for 12 weeks.
  Interventions: Drug: Placebo
- RG7314 (Experimental): Participants will receive RG7314 orally at a dose of 1.5 mg/day in Stage I, 4 mg/day in Stage II, 10 mg/day in Stage III and 1.5 mg/day or 10 mg/day in Stage IV for 12 weeks.
  Interventions: Drug: RG7314

INTERVENTIONS:
Drug: Placebo — Placebo will be administered in different stages of the study for 12 weeks.
  Arms: Placebo
Drug: RG7314 — RG7314 will be administered orally at a dose of 1.5 mg/day in Stage I, 4 mg/day in Stage II, 10 mg/day in Stage III and 1.5 mg/day or 10 mg/day in Stage IV for 12 weeks.
  Arms: RG7314

SUMMARY:
This multi-center, randomized, double-blind, parallel group, placebo-controlled, proof of concept study will investigate the efficacy and safety of RG7314 in adult participants with ASD. In Stage I of the study, participants will be randomized in 2:1 to receive daily oral doses of 1.5 milligrams (mg) RG7314 or placebo for 12 weeks. After an independent safety review, the study may proceed to Stage II. In Stage II of the study, additional participants will be randomized in 2:1 to receive daily oral doses of 4 mg RG7314 or placebo for 12 weeks. After an independent safety review, Stage III will be started wherein additional participants will be randomized in 2:1 to receive daily oral doses of 10 mg RG7314 or placebo for 12 weeks. During Stage III, safety will be reviewed by independent safety review twice and if no safety signal is observed, then additional participants will be randomized in 1:1:1 either to receive 1.5 milligrams per day (mg/day) or 10 mg/day RG7314 orally or placebo for 12 weeks in Stage IV.

ELIGIBILITY:
Inclusion Criteria:

* Participants meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for ASD and Tenth Revision of the International Classification of Diseases and Related Health Problems (ICD-10) criteria for Autism diagnosis
* SRS-2 (T-score) greater than or equal to (>/=) 66
* CGI-S >/=4 (moderately ill)
* Participants have an Intelligence Quotient (IQ) >/=70 (Wechsler Abbreviated State of Intelligence)
* A body mass index (BMI) between 18 to 40 kilograms per square meter (kg/m^2) inclusive
* Language, hearing and vision compatible with the study measurements as judged by the investigator
* Lives with (or has substantial periods of contact with) a caregiver who is willing and able to attend visits when required, oversee the participant's compliance with protocol-specified procedures and study medication dosing, and report on the participant's status via completion of study assessments. Any period of absence must be covered by another caregiver. Non-cohabitating caregiver(s) must spend sufficient time with the participant so that, in the opinion of the investigator, the caregiver(s) can reliably assess participant's mental status, activities and behavior.

Exclusion Criteria:

* Alcohol and/or substance abuse/dependence during the last 12 months
* A significant risk for suicidal behavior, in the opinion of the investigator
* Systolic blood pressure greater than (>) 140 or less than (<) 90 millimeters of mercury (mm Hg), and diastolic blood pressure >90 or less than (<) 50 mm Hg
* Resting pulse rate >90 or <40 beats per minute
* Use of prohibited medications or herbal remedies within 2 weeks prior to randomization, or 5 half-lives (whichever is longer)
* Initiation of a new major change in psychological intervention within 4 weeks prior to randomization. Minor changes in ongoing treatment are not considered significant
* Participation in an investigational drug or device study within 60 days prior to randomization

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 223 (Actual)
Dates: Start 2013-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Social Communication Deficits as Measured by Social Responsiveness Scale 2 (SRS-2) | Baseline, Week 12
Percentage of Participants with Suicidality, as Measured by the Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline up to Week 12
Percentage of Participants With Adverse Events | From Baseline up to Week 18

SECONDARY OUTCOMES:
Change From Baseline in Behavior/Symptoms as Measured by Aberrant Behavior Checklist (ABC) | Baseline, Week 12
Change From Baseline in Behavior/Symptoms as Measured by Repetitive Behavior Scale-Revised (RBS-R) | Baseline, Week 12
Change From Baseline in Behavior/Symptoms as Measured by Anxiety, Depression and Mood Scale (ADAMS) | Baseline, Week 12
Measure: Change From Baseline in Behavior/Symptoms as Measured by State-Trait Anxiety Inventory (STAI) | Baseline, Week 12
Change From Baseline in Clinical Global Impressions as Measured by Clinical Global Impressions Improvement (CGI-I) Scale | Baseline, Week 12
Change From Baseline in Adaptive Functioning and Skills as Measured by Vineland-II Adaptive Behavior Scale (VABS) | Baseline, Week 12
Plasma Concentration of RG7314 | Pre-dose (0 hours [hr]), and 2, 4, 6 hrs post-dose on Day 1, 14, 84; pre-dose (0 hr) on Day 42; any time during early withdrawal visit (up to Week 12)
Plasma Concentration of RG7314 Metabolite M3 | Pre-dose (0 hr), and 2, 4, 6 hrs post-dose on Day 1, 14, 84; pre-dose (0 hr) on Day 42; any time during early withdrawal visit (up to Week 12)
Area Under the Plasma Concentration Versus Time Curve From Time Zero to Last Measurable Concentration (AUClast) of RG7314 | Pre-dose (0 hr), and 2, 4, 6 hrs post-dose on Day 1, 14, 84; pre-dose (0 hr) on Day 42; any time during early withdrawal visit (up to Week 12)
AUClast of RG7314 Metabolite M3 | Pre-dose (0 hr), and 2, 4, 6 hrs post-dose on Day 1, 14, 84; pre-dose (0 hr) on Day 42; any time during early withdrawal visit (up to Week 12)
Maximum Observed Plasma Concentration (Cmax) of RG7314 | Pre-dose (0 hr), and 2, 4, 6 hrs post-dose on Day 1, 14, 84; pre-dose (0 hr) on Day 42; any time during early withdrawal visit (up to Week 12)
Cmax of RG7314 Metabolite M3 | Pre-dose (0 hr), and 2, 4, 6 hrs post-dose on Day 1, 14, 84; pre-dose (0 hr) on Day 42; any time during early withdrawal visit (up to Week 12)
Percentage of Participants With Clinical Response, Defined as At Least 25% Improvement in the SRS-2 Score With a CGI-I Score of 1 or 2 | From Baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (56):
- United States (56):
  - Southwest Autism Research & Resource Center, Phoenix, Arizona
  - Phoenix, Arizona
  - University of California Davis, Sacramento, California
  - Sacramento, California
  - PCSD Feighner Research, San Diego, California
  - San Diego, California
  - University of California at San Francisco, San Francisco, California
  - San Francisco, California
  - Santa Ana, California
  - Stanford, California
  - DBA IMMUNOe Int'l Res Center, Centennial, Colorado
  - Centennial, Colorado
  - Yale University; Yale Child Study Center, New Haven, Connecticut
  - New Haven, Connecticut
  - Neurology offices of south florida, Delray Beach, Florida
  - Delray Beach, Florida
  - Research Centers of America, LLC, Oakland Park, Florida
  - Oakland Park, Florida
  - Compass Research, Orlando, Florida
  - Orlando, Florida
  - Emory University School of Medicine; Department of Human Genetics & Pediatrics, Decatur, Georgia
  - Decatur, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Chicago, Illinois
  - The Kennedy Krieger Institute, Baltimore, Maryland
  - Baltimore, Maryland
  - Neuroscientific Insights, Rockville, Maryland
  - Rockville, Maryland
  - Massachusetts General Hospital, Lexington, Massachusetts
  - Lexington, Massachusetts
  - University of Minnesota; Clin. Neuro Research Unit, Minneapolis, Minnesota
  - Minneapolis, Minnesota
  - Mount Sinai School of Medicine; Seaver Autism Center, New York, New York
  - New York, New York
  - Nathan S. Kline Institute for Psychiatric Research, Orangeburg, New York
  - Orangeburg, New York
  - Montefiore Medical Center; Departments of Psychiatry & Biobehavioral Science, The Bronx, New York
  - The Bronx, New York
  - DUKE SCHOOL OF MEDICINE;Duke Center for Autism and Brain Development, Durham, North Carolina
  - Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cincinnati, Ohio
  - University Hospitals, Cleveland, Ohio
  - Cleveland, Ohio
  - UPMC Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Nashville, Tennessee
  - Road Runner Research, San Antonio, Texas
  - San Antonio, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - Bellevue, Washington
  - Pacific Institute of Medical Sciences, Bothell, Washington
  - Bothell, Washington
  - Seattle Children's Research Institute, Seattle, Washington
  - Seattle, Washington

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711